CLINICAL TRIAL: NCT05840133
Title: The First Affliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Brief Title: Study of Long Non-coding RNA SNHG15 as a Novel Biomarker in HBV Associated HCC
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, ChunqingWang, Intermediate technician, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2023
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: HCC
Keywords: HBV related HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Paired tumor, adjacent non-tumor liver tissues and blood samples from a cohort of HBV-related HCC patients, and blood samples from healthy subjects were selected as control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HBV-associated HCC group: The age and gender of patients are not limited. The patient was finally diagnosed as HBV-associated HCC by imaging examination and pathology.
  Interventions: Diagnostic Test: No intervention was required for patients or control group in this study
- negative control group: The age and sex of this group were matched with that of HBV-associated HCC patient group. The patient did not have any tumor but had HBV infection. The functions of the renal and heart were normal.
  Interventions: Diagnostic Test: No intervention was required for patients or control group in this study
- Healthy control group: The age and sex of the healthy control group were matched with that of HBV-associated HCC patient group. There was no tumor in the liver or other parts of the body, and no tumor in the blood system. The healthy control group did not have any liver benign diseases. There are no inflammatory diseases in other parts of the body. The functions of the liver, kidney, and heart were normal.
  Interventions: Diagnostic Test: No intervention was required for patients or control group in this study

INTERVENTIONS:
Diagnostic Test: No intervention was required for patients or control group in this study — The patient was treated normally and no intervention was required in this study

SUMMARY:
In this study, the investigators will detect the expression of HBV-related HCC biomarker lncRNA SNHG15 in tumor tissues and peripheral blood, to explore the specific molecular markers for the early diagnosis of HBV-related HCC.

DETAILED DESCRIPTION:
Paired hepatitis B virus (HBV)-related hepatocellular carcinoma (HCC) and adjacent liver tissues were selected, and lncRNA SNHG15 was detected by RT-PCR. At the same time, healthy subjects were selected as the control group, and lncRNA SNHG15 in blood was detected by RT-PCR. At the same time, the correlation between lncRNA SNHG15 and the clinical data of patients, such as diagnosis, pathological grading, recurrence, metastasis and survival time was statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The age and sex of the healthy control group were matched with that of HBV-associated patient group. There was no tumor in the other parts of the body, and no tumor in the blood system. The healthy control group did not have any liver benign diseases. There are no inflammatory diseases in other parts of the body; the functions of the liver, kidney, and heart were normal.

Exclusion Criteria:

* The volunteer has tumors in the liver or other parts of the body, or blood system tumors; The volunteer has benign liver diseases; The patient has inflammatory disease elsewhere. If the volunteer has any one of the above diseases, it shall be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No local or systemic treatment was performed before surgery. The patients were finally diagnosed with HBV-related HCC by examination and imaging examination, and the clinicopathologic data were complete.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of lncRNA SNHG15 in HBV-associated HCC patients before surgery | 1 to 3 days before surgery
  The expression of lncRNA SNHG15 in blood samples: The expressions of lncRNA SNHG15 in blood samples were detected by real-time fluorescence quantitative PCR method.

SECONDARY OUTCOMES:
Detection of lncRNA SNHG15 in HBV-associated HCC patients 1 week after surgery | one week after surgery
  1. The expressions of lncRNA SNHG15 in tissues: In the tumor and adjacent tissues from HBV-associated HCC patients, the expressions of lncRNA SNHG15were measured by real-time fluorescence quantitative PCR method.
  2. The expression of lncRNA SNHG15 in blood samples: The expressions of lncRNA SNHG15 in blood samples were detected by real-time fluorescence quantitative PCR method.
Detection of lncRNA SNHG15 in HBV-associated HCC patients at 6 months after surgery | 6 months postoperatively
  The expression of lncRNA SNHG15 in blood samples: The expressions of lncRNA SNHG15 in blood samples were detected by real-time fluorescence quantitative PCR method.
Detection of lncRNA SNHG15 in the control groups as baseline | the level of lncRNA SNHG15 were detected as baseline
  The expression of lncRNA SNHG15 in blood samples: The expressions of lncRNA SNHG15 in blood samples were detected by real-time fluorescence quantitative PCR method.

CONTACTS AND LOCATIONS:
Overall Officials: ChunqingWang [chunqingwang], Dr, Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) until the project is completed. Sharing IPD may be available 1 year after publication.

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Sartorius K, Sartorius B, Aldous C, Govender PS, Madiba TE. Global and country underestimation of hepatocellular carcinoma (HCC) in 2012 and its implications. Cancer Epidemiol. 2015 Jun;39(3):284-90. doi: 10.1016/j.canep.2015.04.006. Epub 2015 Apr 25. PMID 25922178
- [Background] Falade-Nwulia O, Suarez-Cuervo C, Nelson DR, Fried MW, Segal JB, Sulkowski MS. Oral Direct-Acting Agent Therapy for Hepatitis C Virus Infection: A Systematic Review. Ann Intern Med. 2017 May 2;166(9):637-648. doi: 10.7326/M16-2575. Epub 2017 Mar 21. PMID 28319996
- [Background] Polaris Observatory Collaborators. Global prevalence, treatment, and prevention of hepatitis B virus infection in 2016: a modelling study. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):383-403. doi: 10.1016/S2468-1253(18)30056-6. Epub 2018 Mar 27. PMID 29599078
- [Background] Prevention of Infection Related Cancer (PIRCA) Group, Specialized Committee of Cancer Prevention and Control, Chinese Preventive Medicine Association; Non-communicable & Chronic Disease Control and Prevention Society, Chinese Preventive Medicine Association; Health Communication Society, Chinese Preventive Medicine Association. [Strategies of primary prevention of liver cancer in China: expert consensus (2018)]. Zhonghua Yu Fang Yi Xue Za Zhi. 2019 Jan 6;53(1):36-44. doi: 10.3760/cma.j.issn.0253-3766.2018.07.013. Chinese. PMID 30605974
- [Background] Johnson PJ. The role of serum alpha-fetoprotein estimation in the diagnosis and management of hepatocellular carcinoma. Clin Liver Dis. 2001 Feb;5(1):145-59. doi: 10.1016/s1089-3261(05)70158-6. PMID 11218912
- [Background] Befeler AS, Di Bisceglie AM. Hepatocellular carcinoma: diagnosis and treatment. Gastroenterology. 2002 May;122(6):1609-19. doi: 10.1053/gast.2002.33411. PMID 12016426